CLINICAL TRIAL: NCT01016301
Title: Effects of a Clinical Pharmacist Service on Health-related Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Susanna Wallerstedt, MD, PhD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CPS1
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacist service, (Active Comparator): The pharmacist service consists of medication review, drug treatment discussion with the patient, and a medication report.
  Interventions: Other: Pharmacist service
- Control (No Intervention): Usual care

INTERVENTIONS:
Other: Pharmacist service — Medication Review, medication report
  Arms: Pharmacist service,

SUMMARY:
The aim of the present study is to evaluate effects of a clinical pharmacist service on health-related quality of life and prescribing of drugs.

DETAILED DESCRIPTION:
A randomized controlled trial is performed in two internal medicine wards at Sahlgrenska University Hospital, Göteborg, Sweden.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the wards during week days after decision of a ward physician or nurse if the medical condition allows inclusion

Exclusion Criteria:

* Exclusion criteria are poor Swedish language and planned discharge before the intervention can be performed.
* Patients transferred to wards not belonging to the department of medicine or other hospitals during the hospital stay are also excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | 6 months

SECONDARY OUTCOMES:
Prescribing of drugs | Discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Wallerstedt, MD, Ass Prof, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Mölndal, Sweden

REFERENCES:
- [Result] Bladh L, Ottosson E, Karlsson J, Klintberg L, Wallerstedt SM. Effects of a clinical pharmacist service on health-related quality of life and prescribing of drugs: a randomised controlled trial. BMJ Qual Saf. 2011 Sep;20(9):738-46. doi: 10.1136/bmjqs.2009.039693. Epub 2011 Jan 5. PMID 21209140
- [Result] Wallerstedt SM, Bladh L, Ramsberg J. A cost-effectiveness analysis of an in-hospital clinical pharmacist service. BMJ Open. 2012 Jan 5;2(1):e000329. doi: 10.1136/bmjopen-2011-000329. Print 2012. PMID 22223840